CLINICAL TRIAL: NCT00105885
Title: Telephone Care as a Substitute for Routine Psychiatric Medication Management
Brief Title: Telephone Care as a Substitute for Routine Psychiatric Medication
Acronym: Telepsych
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEL 01-146
Record Dates: First submitted 2005-03-17; First posted 2005-03-18 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2008-10

CONDITIONS: Major Depression; Posttraumatic Stress Disorders; Anxiety Disorders
Keywords: Telephone; Telemedicine; Psychopharmacology
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Patients randomized to receive telephone care will be scheduled to see their provider at twice the recommended clinical visit interval, and two ten-minute telephone contacts will be scheduled at a specific time at standard 0.67 and 1.3 times the multiple of the recommended interval.
  Interventions: Procedure: telephone care
- Arm 2 (No Intervention): Patients randomized to receive routine care will be scheduled to see their psychiatric medication provider at the recommended interval.

INTERVENTIONS:
Procedure: telephone care — Patients randomized to receive telephone care will be scheduled to see their provider at twice the recommended clinical visit interval, and two ten-minute telephone contacts will be scheduled at a specific time at standard 0.67 and 1.3 times the multiple of the recommended interval.
  Arms: Arm 1

SUMMARY:
The purpose of this study is to answer the following questions: (1) Does substituting brief, scheduled, clinician-initiated telephone calls (telephone care) for routine psychiatric medication management visits reduce overall healthcare utilization? (2) Is substituting brief, scheduled, clinician-initiated telephone calls (telephone care) for routine psychiatric medication management visits as effective as routine care?

DETAILED DESCRIPTION:
Telemedicine uses communications technologies to provide health care when distance separates participants. Applied to general medical care practice, telemedicine is associated with improved continuity of care, cost-effectiveness, and improved service quality. To date, all evaluations of telepsychiatry have concentrated on video technology. The telephone is more readily available and less expensive communication technology that has not been evaluated as a method of health services delivery in the medication management of stable psychiatric outpatients. We will enroll 346 psychiatrically stable subjects, who carry a diagnosis of major depression, post-traumatic stress disorder (PTSD) or non-PTSD anxiety disorder. We will use a balanced randomization strategy to assign subjects to routine care or telephone care for a two-year period within each provider panel. Patients randomized to receive routine care will be scheduled to see their psychiatric medication provider at the recommended interval. Patients randomized to receive telephone care will be scheduled to see their provider at twice the recommended clinic visit interval, and two ten-minute telephone contacts will be scheduled at a specific time at standard 0.67 and 1.3 times the multiple of the recommended interval. At two years, we will use ten data sources to compare two primary outcomes (total VHA health services utilization and mental health component scores from the SF-12-V) as well as VHA costs, imputed non-VHA costs, patient and provider satisfaction, medication compliance and diagnosis specific outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for this study if they carry a diagnosis of major depression, Post-traumatic Stress Disorder (PTSD), or non-PTSD anxiety disorders.
* They must be psychiatrically stable subjects with a Global Assessment of Functioning scale score of >50, no psychiatric hospitalizations in the previous six months, and no active substance abuse disorders.

Exclusion Criteria:

* Psychiatric hospitalization within 6 months prior to study entry.
* Visit interval >1 year.
* Lack of telephone access.
* Inability to use a telephone.
* GAF<50.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2003-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization (VHA and non-VHA patient visits); patient time spent obtaining care (including travel time); time provider spends in direct patient care. | Continuous

SECONDARY OUTCOMES:
Patient satisfaction at baseline, midpoint, end of study; provider satisfaction at baseline, midpoint, end of study; patient medication compliance; SF12V and brief symptom checklist scores | baseline, 6 months, 12 months, 18 months, 24 months
SF12V and brief symptom checklist scores | baseline, 6 months, 18 months, 24 months
patient medication compliance | two month intervals
provider satisfaction | baseline, midpoint, and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Amy E. Wallace, MD MPH, Principal Investigator — VA Medical & Regional Office Center, White River
Locations (1):
- VA Medical & Regional Office Center, White River, White River Junction, Vermont, United States

REFERENCES:
- [Result] Pomerantz A, Cole BH, Watts BV, Weeks WB. Improving efficiency and access to mental health care: combining integrated care and advanced access. Gen Hosp Psychiatry. 2008 Nov-Dec;30(6):546-51. doi: 10.1016/j.genhosppsych.2008.09.004. Epub 2008 Oct 5. PMID 19061681
- [Result] Morden NE, Mistler LA, Weeks WB, Bartels SJ. Health care for patients with serious mental illness: family medicine's role. J Am Board Fam Med. 2009 Mar-Apr;22(2):187-95. doi: 10.3122/jabfm.2009.02.080059. PMID 19264942